CLINICAL TRIAL: NCT05070000
Title: Value of Ultrasound and Computed Tomography in the Diagnosis of Acute Appendicitis With Histopathology as Gold Standard - Retrospective Cohort Study.
Brief Title: Value of Ultrasound and Computed Tomography in the Diagnosis of Acute Appendicitis With Histopathology as Gold Standard.
Status: Completed | Type: Observational
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Louis Haentjens, M.D, KU Leuven
Other Study IDs: Appendixstudy
Record Dates: First submitted 2021-07-30; First posted 2021-10-06 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: Appendicitis Acute
Keywords: Appendicitis; General Surgery; Ultrasound; Computed Tomography
MeSH Terms: conditions — Appendicitis | interventions — Diagnostic Imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- US: Ultrasound
- CT: Computed tomography
- US after CT: Ultrasound after Computed tomography
  Interventions: Diagnostic Test: Radiologic examination

INTERVENTIONS:
Diagnostic Test: Radiologic examination — Patients underwent US, CT or CT after US
  Groups: US after CT

SUMMARY:
This study is a retrospective evaluation of all patients treated surgically for appendicitis over a period of 3 years at the Sint- Andries Hospital, Tielt. Belgium. The goal is to evaluate the value of ultrasound (US), computed tomography (CT) and laboratory testing in diagnosing acute appendicitis and to look for the possible impact on the treatment.

ELIGIBILITY:
Inclusion Criteria:

* suspicion of acute appendicitis

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients at the emergency departement with clinical signs of acute appendicitis
Sampling Method: Probability Sample
Enrollment: 304 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of diagnostic test | 3 years
  For US and CT sensitivity and specificity for diagnosing acute appendicitis were evaluated.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Marzuillo P, Germani C, Krauss BS, Barbi E. Appendicitis in children less than five years old: A challenge for the general practitioner. World J Clin Pediatr. 2015 May 8;4(2):19-24. doi: 10.5409/wjcp.v4.i2.19. eCollection 2015 May 8. PMID 26015876
- [Background] Shogilev DJ, Duus N, Odom SR, Shapiro NI. Diagnosing appendicitis: evidence-based review of the diagnostic approach in 2014. West J Emerg Med. 2014 Nov;15(7):859-71. doi: 10.5811/westjem.2014.9.21568. Epub 2014 Oct 7. PMID 25493136
- [Background] Drake FT, Flum DR. Improvement in the diagnosis of appendicitis. Adv Surg. 2013;47:299-328. doi: 10.1016/j.yasu.2013.03.003. PMID 24298858
- [Background] Drake FT, Mottey NE, Farrokhi ET, Florence MG, Johnson MG, Mock C, Steele SR, Thirlby RC, Flum DR. Time to appendectomy and risk of perforation in acute appendicitis. JAMA Surg. 2014 Aug;149(8):837-44. doi: 10.1001/jamasurg.2014.77. PMID 24990687
- [Result] Eng KA, Abadeh A, Ligocki C, Lee YK, Moineddin R, Adams-Webber T, Schuh S, Doria AS. Acute Appendicitis: A Meta-Analysis of the Diagnostic Accuracy of US, CT, and MRI as Second-Line Imaging Tests after an Initial US. Radiology. 2018 Sep;288(3):717-727. doi: 10.1148/radiol.2018180318. Epub 2018 Jun 19. PMID 29916776
- [Result] Weston AR, Jackson TJ, Blamey S. Diagnosis of appendicitis in adults by ultrasonography or computed tomography: a systematic review and meta-analysis. Int J Technol Assess Health Care. 2005 Summer;21(3):368-79. doi: 10.1017/s0266462305050488. PMID 16110717
- [Result] Johansson EP, Rydh A, Riklund KA. Ultrasound, computed tomography, and laboratory findings in the diagnosis of appendicitis. Acta Radiol. 2007 Apr;48(3):267-73. doi: 10.1080/02841850601182162. PMID 17453494
- [Result] Khan MN, Davie E, Irshad K. The role of white cell count and C-reactive protein in the diagnosis of acute appendicitis. J Ayub Med Coll Abbottabad. 2004 Jul-Sep;16(3):17-9. PMID 15631364
- [Result] McGowan DR, Sims HM, Zia K, Uheba M, Shaikh IA. The value of biochemical markers in predicting a perforation in acute appendicitis. ANZ J Surg. 2013 Jan;83(1-2):79-83. doi: 10.1111/ans.12032. Epub 2012 Dec 12. PMID 23231057
- [Result] Meltzer AC, Baumann BM, Chen EH, Shofer FS, Mills AM. Poor sensitivity of a modified Alvarado score in adults with suspected appendicitis. Ann Emerg Med. 2013 Aug;62(2):126-31. doi: 10.1016/j.annemergmed.2013.01.021. Epub 2013 Apr 24. PMID 23623557
- [Result] Luckmann R, Davis P. The epidemiology of acute appendicitis in California: racial, gender, and seasonal variation. Epidemiology. 1991 Sep;2(5):323-30. doi: 10.1097/00001648-199109000-00003. PMID 1742380
- [Result] Kaiser S, Mesas-Burgos C, Soderman E, Frenckner B. Appendicitis in children--impact of US and CT on the negative appendectomy rate. Eur J Pediatr Surg. 2004 Aug;14(4):260-4. doi: 10.1055/s-2004-817841. PMID 15343467